CLINICAL TRIAL: NCT02740816
Title: Comparative Study of Menstrual Blood and Systemic Blood: Quantifying the Difference
Brief Title: Comparative Study of Menstrual Blood and Systemic Blood
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul D Blumenthal, Professor, Stanford University
Other Study IDs: 35817
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Retention; Menstruation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Menstrual Blood and Systemic Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Comparative blood analysis — Collection of menstrual blood and systemic blood

SUMMARY:
The purpose is to investigate how menstrual blood differs from systemic blood to evaluate if menstrual blood could be utilized as a natural and non-invasive access to blood for regular health monitoring and early diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45

Exclusion Criteria:

* weigh less then 110 pounds
* currently on a birth control method

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy menstruating women.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Health Markers in Systemic Blood vs. Menstrual Blood | Up to 2 months
  The following biomarkers will be tested for and then compared for systemic blood and menstrual blood:
  * BUN
  * Sodium
  * Potassium
  * Chloride
  * Glucose
  * Calcium
  * HDL
  * LDL
  * Triglycerides
  * CRP
  * Estradiol
  * Ferritin
  * A1c
  * Hemoglobin
  * Hepatic function panel
  * TSH
  * FSH
  * T3

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Blumenthal, MD, MPH, Principal Investigator — Stanford University, Department of OB/GYN
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No